CLINICAL TRIAL: NCT05251116
Title: Accuracy Study of an Interstitial Fluid Glucose Sensor
Brief Title: Study of an Interstitial Fluid Glucose Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADC-US-VAL-21206
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- only one Arm is included in this study (Other): This is a non-randomized, single arm study. All subjects will use the System. Results from the System will be compared to reference instrument.
  Interventions: Device: FreeStyle Libre

INTERVENTIONS:
Device: FreeStyle Libre — FreeStyle Libre 2 continuous Glucose Monitoring System

SUMMARY:
To characterize the System performance with respect to Yellow Springs Instrument (YSI) reference venous plasma measurements. Safety of the investigational device will be characterized by Adverse Device Effects and Serious Adverse Device Effects experienced by study participants.

DETAILED DESCRIPTION:
Up to 200 adult and 250 pediatric (17 years of age or younger) subjects will be enrolled to obtain at least 200 evaluable subjects. At least four (4) subjects between the ages of 2 and 5 will be enrolled. Subjects will wear a total of two (2) sensors, one on the back of each upper arm.

Each subject will wear two sensors, from the same Sensor lot, one on the back of each upper arm. One or more unique sensor lots will be evaluated in this study. Subjects will make between four (4) and six (6) scheduled visits to the clinical study site, including the Enrollment/Screening Visit (Visit 1). Subjects aged 2 - 5 will have one (1) in-clinic visit where capillary blood testing will be performed. Based on the subjects age and/or weight, subjects age 6 or older, will have up to three in-clinic visits during which intravenous blood draws and YSI reference testing will occur. Based on the subjects' age, blood glucose levels may be manipulated.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be considered eligible for participation in the study:

1. Subject must be at least 2 years of age.
2. Subject must have type 1 or type 2 diabetes.
3. Subject must require insulin therapy through an insulin pump and/or multiple daily insulin injections (at least 3 injections daily).
4. Willing to perform a minimum of 4 finger sticks per day while wearing the sensor in the study.
5. Subject and/or guardian must be able to read and understand English.
6. For subjects age between 2 and 5: willing to allow medical personnel to perform up to 16 capillary finger sticks to allow for capillary blood samples to be obtained per the study protocol.
7. For subjects age 6 and older: willing to allow medical personnel to insert an IV catheter in the arm to allow for venous blood samples to be obtained per the study protocol.
8. For subjects age 11 and older: subject is willing to have their blood sugar manipulated during one or more in-clinic sessions.
9. In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
10. At the time of enrollment, subject must be available to participate in all study visits.
11. Known insulin sensitivity factor (only applicable to subjects age 11 and older)
12. Subjects aged 18 years and older must be willing and able to provide written signed and dated informed consent.
13. Subjects aged 17 years and younger must have a parent, guardian or legally authorized representative willing and able to provide written informed consent.
14. Subjects aged 7 - 17 years of age must be willing and able to provide written signed and dated informed assent.

    Exclusion Criteria:

    Subjects must not meet exclusion criteria to be considered eligible for participation in the study. The subject will be excluded from the study if:
15. Subject has a history of hypoglycemia unawareness (only applicable to subjects age 11 and older).
16. Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
17. Subjects age 11 and older: Subject is known to be pregnant, attempting to conceive or is not willing and able to practice birth control during the study duration (applicable to only to female subjects age 11 and older).
18. Subjects age 10 and younger: Subject is known to be pregnant or becomes pregnant during the study (only applicable to female subjects age 10 years and younger)
19. Subject has extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements. Such conditions include, but are not limited to extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, dermatitis herpetiformis, skin lesions, redness, infection or edema.
20. Subject has had an episode of severe hypoglycemia requiring intervention from a health care professional (i.e. EMT assistance, emergency room visit, or hospital admission) within the last six (6) months (only applicable to subjects age 11 and older).
21. Subject has had an episode of diabetic ketoacidosis (DKA) within the last three (3) months (only applicable to subjects age 11 and older).
22. Subject is currently participating in another clinical trial.
23. Subject has donated blood within 112 days (3.7 months) prior to the beginning of the study activities.
24. For subjects age 6 and older: subject has a hemoglobin (Hb) level that is below the normal range (for reference the low end of the normal range for Hb for adult males is 14 g/dL and for adult females is 12 g/dL1; for pediatric males and pediatric females aged 6 - 12 years old it is 11.5 g/dL; for pediatric males aged 12 - 17 it is 13.0 g/dL; for pediatric females aged 12 - 17 it is 12.0 g/dL2).
25. Subject has a known concomitant medical condition which, in the opinion of the investigator, could present a risk to the safety or welfare of the subject or study staff.
26. Subject has X-ray, MRI, CT or diathermy appointment scheduled during the period of study participation, and the appointment cannot be rescheduled for a time before study participation starts or after study participation ends.
27. Subject is unsuitable for participation due to any other cause as determined by the investigator.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2021-12-11 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
System Performance | 46 Days
  System Performance will be evaluated against the reference system, Yellowstone Instrument (YSI) and against Capillary blood Glucose (BG). During several in clinic visits, plasma samples obtained from the subjects at various time intervals will be analyzed using the YSI. Results will be compared with results obtained from the System, to determine the system accuracy. Similarly, capillary Blood Glucose will be measured and compared with results obtained from the system.

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara A Karinka, PhD, Study Director — Abbott Diabetes Care
Locations (5):
- United States (5):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rocky Mountain Diabetes & Osteoporosis Center, Idaho Falls, Idaho
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas
  - Rainier Clinical Research, Renton, Washington

IPD SHARING:
Plan to Share IPD: No